CLINICAL TRIAL: NCT04585789
Title: A Phase 2 Randomized, Open-label, Parallel-group, Multicenter Study to Assess Intrahepatic and Peripheral Changes of Immunologic and Virologic Markers in Response to Combination Regimens Containing JNJ-73763989 and Nucleos(t)Ide Analog With or Without JNJ-56136379 in Patients With Chronic Hepatitis B Virus Infection
Brief Title: A Study to Assess Intrahepatic and Peripheral Changes of Immunologic and Virologic Markers in Chronic Hepatitis B Virus Infection
Acronym: INSIGHT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CR108790; 73763989HPB2003 (Other: Janssen Research & Development, LLC); 2019-004475-39 (EudraCT Number)
Record Dates: First submitted 2020-10-09; First posted 2020-10-14 (Actual); Results first posted 2024-03-05 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — JNJ-56136379; entecavir; Tenofovir; tenofovir alafenamide

STUDY DESIGN:
Intervention Model Description: As per protocol amendment-5, JNJ-56136379 has been removed as study intervention and all participants are counted as single arm in each panel.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Panel 1: JNJ-73763989+ NA (Experimental): Ongoing and new participants will receive JNJ-73763989 subcutaneous (SC) injection once every 4 weeks (last injection at Week 44) and nucleos(t)ide analog (NA) treatment (either entecavir [ETV], tenofovir disoproxil or tenofovir alafenamide [TAF] tablets) once daily up to 48 weeks. Participants may receive optional treatment with pegylated interferon alpha-2a (PegIFN-alpha-2a) after the Week 40 for a duration of either 12 or 24 weeks at the investigator's discretion. As per amendment-5, JNJ-56136379 is no longer included as part of the study intervention and all participants are counted as single arm in each panel.
  Interventions: Drug: JNJ-73763989; Drug: JNJ-56136379; Drug: Entecavir (ETV); Drug: Tenofovir disoproxil; Drug: Tenofovir alafenamide (TAF); Drug: PegIFN-alpha-2a (Optional)
- Panel 2: JNJ-73763989+ NA (Experimental): Ongoing and new participants will receive JNJ-73763989 SC injection once every 4 weeks (last injection at Week 44) and NA treatment (ETV, tenofovir disoproxil or TAF tablets) once daily up to 48 weeks. Participants may receive optional treatment with PegIFN-alpha-2a after the Week 40 for a duration of either 12 or 24 weeks at the investigator's discretion. As per amendment-5, JNJ-56136379 is no longer included as part of the study intervention and all participants are counted as single arm in each panel.
  Interventions: Drug: JNJ-73763989; Drug: JNJ-56136379; Drug: Entecavir (ETV); Drug: Tenofovir disoproxil; Drug: Tenofovir alafenamide (TAF); Drug: PegIFN-alpha-2a (Optional)

INTERVENTIONS:
Drug: JNJ-73763989 — JNJ-73763989 will be administered subcutaneously once every 4 weeks up to Week 44.
Drug: JNJ-56136379 — JNJ-56136379 tablets will be administered orally once daily up to 48 weeks.
Drug: Entecavir (ETV) — ETV tablet will be administered orally once daily up to 48 weeks as NA treatment.
Drug: Tenofovir disoproxil — Tenofovir disoproxil will be administered orally once daily up to 48 weeks as NA treatment.
Drug: Tenofovir alafenamide (TAF) — TAF will be administered orally once daily up to 48 weeks as NA treatment.
Drug: PegIFN-alpha-2a (Optional) — PegIFN-alpha-2a injection will be administered subcutaneously once weekly after Week 40 for either 12 or 24 weeks.

SUMMARY:
The purpose of this study is to assess changes in intrahepatic hepatitis B surface antigen (HBsAg) between baseline and on-treatment liver biopsy in response to JNJ-3989-based combination treatment.

DETAILED DESCRIPTION:
The title of protocol reflects the original study design. The study design section is reflecting that the design as of protocol amendment 5 is non-randomized.

ELIGIBILITY:
Inclusion Criteria:

* Medically stable on the basis of physical examination, medical history, vital signs, and triplicate 12-lead electrocardiogram (ECG) performed at screening
* Hepatitis B virus (HBV) infection with documentation at least 6 months prior to screening: participants be either currently not treated with HBeAg positive status or virologically (nucleos[t]ide analog [NA]) suppressed with HBeAg negative status
* Hepatitis B surface antigen (HBsAg) greater than (>) 100 International Units per Milliliter (IU/mL) at screening
* Body mass index (BMI) between 18.0 and 35.0 kilogram per meter square (kg/m^2), extremes included
* Highly effective contraceptive measures in place for female participants of childbearing potential or male participants with female partners of childbearing potential
* Fibroscan liver stiffness measurement less than and equal to (<=) 9 Kilopascal (kPa) within 6 months prior to screening or at the time of screening

Exclusion Criteria:

* Evidence of infection with hepatitis A, C, D or E virus infection or evidence of human immunodeficiency, virus type 1 (HIV-1) or HIV-2 infection at screening
* History or evidence of clinical signs/symptoms of hepatic decompensation including but not limited to: portal hypertension, ascites, hepatic encephalopathy, esophageal varices
* History or signs of cirrhosis or portal hypertension, signs of hepatocellular carcinoma (HCC) or clinically relevant renal abnormalities on an abdominal ultrasound performed within 6 months prior to screening or at the time of screening
* Presence of coagulopathy or bleeding disorder as indicated by: (a) International normalized ratio (INR) greater than or equal to (>=) 1.1* upper limit of normal (ULN); (b) Partial thromboplastin time >1.1*ULN; (c) Any signs of prolonged bleeding (>10 minutes)
* Presence of hemoglobinopathy (including sickle cell disease, thalassemia)
* Liver biopsy performed prior to screening that led to complications and that in the opinion of the investigator would prohibit another liver biopsy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2023-02-08 (Actual); Study Completion 2024-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (10):
- Johns Hopkins University, Baltimore, Maryland, United States
- UZ Antwerpen, Edegem, Belgium
- Toronto General Hospital, Toronto, Ontario, Canada
- Hopital Beaujon, Clichy, France
- University Medical Center, Hamburg, Germany
- Irccs Ospedale Maggiore Di Milano, Milan, Italy
- New Zealand Clinical Research, Auckland, New Zealand
- ID Clinic, Mysłowice, Poland
- United Kingdom (2):
  - Grahame Hayton Unit, London
  - Kings College Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study consisted of 3 Panels (1, 2 and 3). Panel 1: participants with hepatitis B (HB) e antigen (HBeAg) positive and not treated. Panel 2: participants with HBeAg negative and virologically suppressed by entecavir (ETV), tenofovir disoproxil (TD), or tenofovir alafenamide (TAF) treatment. Panel 3: participants with HBeAg positive or negative who were either not treated or virologically suppressed by ETV or TD treatment.
Pre-assignment Details: As per protocol amendment (PA) 5 (dated 01 October 2021), all participants stopped JNJ-56136379 (JNJ-6379) treatment and continued treatment with JNJ-73763989 (JNJ-3989) plus nucleos(t)ide analog (NA; ETV, TD, or TAF) plus optional pegylated interferon alpha-2a (PegIFN-alpha2a). The study consisted of 3 phases: screening phase, open-label (OL) intervention phase and follow-up (FU) phase.
Groups:
- Panel 1: Prior to PA 5, participants received either JNJ-3989 200 milligrams (mg) subcutaneous(SC) injection every 4 weeks(Q4W) from Day 1 (Week 1) to Week 44+JNJ-6379 250 mg once daily(QD)+NA (ETV 0.5 mg/TD 245 mg/TAF 25 mg) QD from Day 1 (Week 1) to Week 48 or JNJ-3989 200 mg SC injection Q4W from Day 1 (Week 1) to Week 44+NA (ETV 0.5 mg/TD 245 mg/TAF 25 mg) QD from Day 1 (Week 1) to Week 48. After PA 5, participants stopped JNJ-6379 and continued JNJ-3989+NA. With separate consent, participants received optional treatment:PegIFN-alpha-2a 180 micrograms(mcg) SC injection once weekly(QW) post Week 40 liver biopsy for either 12/24 weeks (anytime between study Week 40 to 72) at investigator's discretion. At end of treatment Week 48, all participants entered FU phase; stopped JNJ-3989/JNJ-6379 and NA ( if NA completion criteria [NAcc:alanine aminotransferase {ALT} less than {<}3*upper limit of normal{ULN}, HB virus deoxyribonucleic acid {HBV DNA} <lower limit of quantification {LLOQ}:20 International Units per milliliter {IU/mL}], HBeAg negative & HB surface antigen {HBsAg} <10 IU/mL] was met as per Week 44 laboratory tests). If NAcc were not met, NA was continued till FU end (study Week 96). Participants on PegIN-alpha2a and who had not met NAcc at Week 48 were assessed at PegIN-alpha2a treatment end and stopped NA, if NAcc was met; then entered FU. If NA-retreatment criteria (HBV DNA >20,000 IU/mL, HBV DNA >2,000 IU/mL but <20,000 IU/mL & ALT >5*ULN) was met in FU, NA was re-started.
- Panel 2: Prior to PA 5, participants received either JNJ-3989 200 mg SC injection Q4W from Day 1 (Week 1) to Week 44 + JNJ-6379 250 mg QD and NA treatment (ETV 0.5 mg/TD 245 mg/TAF 25 mg) QD from Day 1 (Week 1) to Week 48, or JNJ-3989 200 mg SC injection Q4W from Day 1 (Week 1) to Week 44 + NA (ETV 0.5 mg/TD 245 mg/TAF 25 mg) QD from Day 1 (Week 1) to Week 48. After PA 5, participants discontinued JNJ-6379 and continued JNJ-3989 + NA. With separate consent, participants received optional treatment with PegIFN-alpha-2a 180 mcg SC injection QW after Week 40 liver biopsy for either 12 or 24 weeks (anytime between study Week 40 to 72) at investigator's discretion. At end of treatment Week 48, all participants entered FU phase and stopped JNJ-3989/JNJ-6379 and NA (if NA treatment completion criteria [ALT <3*ULN, HBV DNA <LLOQ; 20 IU/mL, HBeAg negative and HBsAg <10 IU/mL] was met as per Week 44 laboratory tests). If NA completion criteria were not met, NA was continued till FU phase end (study Week 96). Participants on PegIN-alpha2a and who had not met NA completion criteria at Week 48 were assessed at end of PegIN-alpha2a treatment and stopped NA, if completion criteria met and then entered FU phase. If NA-retreatment criteria (HBV DNA >20,000 IU/mL, HBV DNA >2,000 IU/mL but <20,000 IU/mL and ALT >5*ULN) were met in FU phase, NA retreatment was started.
- Panel 3: After PA 5, participants received JNJ-3989 200 mg SC injection Q4W from Day 1 (Week 1) to Week 44 + NA treatment (ETV 0.5 mg/TD 245 mg/TAF 25 mg) QD from Day 1 (Week 1) to Week 48. With separate consent, participants received optional treatment with PegIFN-alpha-2a 180 mcg SC injection QW after Week 40 liver biopsy for either 12 or 24 weeks (anytime between study Week 40 to 72) at investigator's discretion. At end of treatment Week 48, all participants entered follow-up and stopped JNJ-3989 and NA (if NA treatment completion criteria [ALT <3*ULN, HBV DNA <LLOQ; 20 IU/mL, HBeAg negative and HBsAg <10 IU/mL] was met based on Week 44 laboratory tests). If NA completion criteria were not met, NA was continued till FU phase end (study Week 96). Participants on PegIN-alpha2a and who had not met NA completion criteria at Week 48 were assessed at end of PegIN-alpha2a treatment and stopped NA, if completion criteria met and then entered FU phase. If NA-retreatment criteria (HBV DNA >20,000 IU/mL, HBV DNA >2,000 IU/mL but <20,000 IU/mL and ALT >5*ULN) were met in FU phase, NA retreatment was started.
Period: OL Phase: Week 1 to Week 48
Arm/Group | Panel 1 | Panel 2 | Panel 3
Started | 10 | 10 | 4
Completed | 10 | 10 | 4
Not Completed | 0 | 0 | 0
Period: FU Phase: Week 48 to Week 96
Arm/Group | Panel 1 | Panel 2 | Panel 3
Started | 10 | 10 | 4
Completed | 8 | 10 | 4
Not Completed | 2 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Panel 1 | Panel 2 | Panel 3 | Total
Number analyzed (Participants) | 10 | 10 | 4 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.4 (14.73) | 43.4 (12.63) | 42 (12.73) | 39 (13.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 0 | 10
  Male | 5 | 5 | 4 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 10 | 9 | 4 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 8 | 3 | 0 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 3 | 7
  White | 0 | 4 | 1 | 5
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  BELGIUM | 1 | 1 | 0 | 2
  CANADA | 5 | 0 | 0 | 5
  FRANCE | 0 | 1 | 4 | 5
  GERMANY | 0 | 1 | 0 | 1
  ITALY | 3 | 2 | 0 | 5
  NEW ZEALAND | 1 | 2 | 0 | 3
  POLAND | 0 | 1 | 0 | 1
  UNITED KINGDOM | 0 | 1 | 0 | 1
  UNITED STATES | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Panel 1 and 2: Absolute Change From Baseline in the Percentage of Hepatitis B Surface Antigen (HBsAg) Hepatocytes at Week 40
Description: Absolute change from baseline to on-treatment liver biopsy timepoint (Week 40) in terms of the percentage of HBsAg-positive hepatocytes (at Week 40) were reported.
Time Frame: Baseline, Week 40
Population: Intent-to-treat (ITT) population included participants who were randomly assigned or enrolled to an intervention arm and received at least 1 dose of intervention. Participants were analyzed according to study intervention they were randomly assigned or enrolled. Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure. Data for this outcome measure was planned to be collected and analyzed for Panels 1 and 2 alone.
Measure: Mean (80% Confidence Interval); unit: percentage of HBsAg hepatocytes
Arm/Group | Panel 1 | Panel 2
Number analyzed (Participants) | 6 | 9
percentage of HBsAg hepatocytes | -78.46 [-94.078 to -42.936] | -5.68 [-15.846 to -0.885]

2. Primary Outcome: Panel 3: Liver Concentrations of JNJ-73763989 (JNJ-73763976, JNJ-73763924 and JNJ-87719164 [M65; Deaminated Metabolite of JNJ-73763976]) at Week 12
Description: Liver concentrations of JNJ-73763989 (JNJ-73763976, JNJ-73763924 - Molecules of JNJ-73763989 and JNJ-87719164 [M65; deaminated metabolite of JNJ-73763976]) at Week 12 were reported.
Time Frame: At Week 12 (at the time of liver biopsy: 24 hours post dose of JNJ-73763989)
Population: ITT population included participants who were randomly assigned or enrolled to an intervention arm and received at least 1 dose of intervention. Participants were analyzed according to study intervention they were randomly assigned or enrolled. Data for this outcome measure was planned to be collected and analyzed for Panel 3 alone.
Measure: Mean (Standard Deviation); unit: nanograms per gram (ng/g)
Arm/Group | Panel 3
Number analyzed (Participants) | 4
nanograms per gram (ng/g)
  JNJ-73763976 | 3550.00 (1674.714)
  JNJ-73763924 | 87300.00 (31712.668)
  M65 | 66175.00 (26000.817)

3. Primary Outcome: Panel 3: Liver Concentrations of JNJ-73763989 (JNJ-73763976, and JNJ-73763924 and JNJ-87719164 [M65; Deaminated Metabolite of JNJ-73763976]) at Week 40
Description: Liver concentrations of JNJ-73763989 (JNJ-73763976, and JNJ-73763924 and JNJ-87719164 [M65; deaminated metabolite of JNJ-73763976]) at Week 40 were reported.
Time Frame: At Week 40 (at the time of liver biopsy: 24 hours post dose of JNJ-73763989)
Population: ITT population included participants who were randomly assigned or enrolled to an intervention arm and received at least 1 dose of intervention. Participants were analyzed according to study intervention they were randomly assigned or enrolled. Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure. Data for this outcome measure was planned to be collected and analyzed for Panel 3 alone.
Measure: Mean (Standard Deviation); unit: ng/g
Arm/Group | Panel 3
Number analyzed (Participants) | 3
ng/g
  JNJ-73763976 | 5883.33 (2147.145)
  JNJ-73763924 | 208666.67 (66860.551)
  M65 | 133800.00 (50615.413)

4. Primary Outcome: Panel 3: Plasma Concentration of JNJ-73763989 (JNJ-73763976, and JNJ-73763924) at Week 12
Description: Plasma concentration of JNJ-73763989 (JNJ-73763976 and JNJ-73763924-molecules of JNJ-73763989) at Week 12 were reported.
Time Frame: At Week 12 (at the time of liver biopsy: 24 hours post dose of JNJ-73763989)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nanograms per milliliters (ng/mL)
Arm/Group | Panel 3
Number analyzed (Participants) | 4
nanograms per milliliters (ng/mL)
  JNJ-73763976 | 254.70 (123.841)
  JNJ-73763924 | 36.18 (22.667)

5. Primary Outcome: Panel 3: Plasma Concentrations of JNJ-73763989 (JNJ-73763976 and JNJ-73763924) at Week 40
Description: Plasma concentrations of JNJ-73763989 (JNJ-73763976 and JNJ-73763924-molecules of JNJ-73763989) at Week 40 were reported.
Time Frame: At Week 40 (at the time of liver biopsy: 24 hours post dose of JNJ-73763989)
Population: ITT population included participants who were randomly assigned or enrolled to an intervention arm and received at least 1 dose of intervention. Participants were analyzed according to study intervention they were randomly assigned or enrolled. Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure. Data for this outcome measure (OM) was planned to be collected and analyzed for Panel 3 alone.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Panel 3
Number analyzed (Participants) | 3
ng/mL
  JNJ-73763976 | 530.97 (176.408)
  JNJ-73763924 | 74.87 (12.788)

6. Primary Outcome: Panel 3: Correlation of Liver Concentration to Plasma Concentration of JNJ-73763989 (JNJ-73763976 and JNJ-73763924) and Liver Concentration of JNJ-87719164 (M65: Deaminated Metabolite of JNJ-73763976) to Liver Concentration JNJ-73763976 at Week 12
Description: Correlation of liver concentration to plasma concentration of JNJ-73763989 (JNJ-73763976 and JNJ-73763924) and liver concentration of JNJ-87719164 (M65: Deaminated metabolite of JNJ-73763976) to liver concentration JNJ-73763976 at Week 12 were reported.
Time Frame: Week 12 (at the time of liver biopsy: 24 hours post dose of JNJ-73763989)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Panel 3
Number analyzed (Participants) | 4
ratio
  JNJ-73763976 (liver to plasma concentration) | 14.51 (4.725)
  JNJ-73763924 (liver to plasma concentration) | 2844.26 (1265.202)
  M65 to JNJ-73763976 (liver to liver concentration) | 19.47 (3.267)

7. Primary Outcome: Panel 3: Correlation of Liver to Plasma Concentration of JNJ-73763989 (JNJ-73763976 and JNJ-73763924) and Liver Concentration of JNJ-87719164 (M65: Deaminated Metabolite of JNJ-73763976) to Liver Concentration JNJ-73763976 at Week 40
Description: Correlation of liver concentration to plasma concentration of JNJ-73763989 (JNJ-73763976 and JNJ-73763924) and liver concentration of JNJ-87719164 (M65: Deaminated metabolite of JNJ-73763976) to liver concentration JNJ-73763976 at Week 40 were reported.
Time Frame: Week 40 (at the time of liver biopsy: 24 hours post dose of JNJ-73763989)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Panel 3
Number analyzed (Participants) | 3
ratio
  JNJ-73763976 (liver to plasma concentration) | 12.67 (7.269)
  JNJ-73763924 (liver to plasma concentration) | 2847.66 (1034.033)
  M65 to JNJ-73763976 (liver to liver concentration) | 22.65 (1.407)

8. Secondary Outcome: Panel 1, 2 and 3: Percentage of Participants With Sustained (Reduction) Serum HBsAg Response Per Definition 2 at Follow-up Week 48
Description: Percentage of participants with sustained (reduction) serum HBsAg response per Definition 2 at follow-up Week 48 were reported. Sustained serum HBsAg response per definition 2 was defined as: for participants with a >1 log decline in HBsAg from baseline at last follow up visit: Among the most recent three visits, the difference between log HBsAg at 2 of 3 last visit and 1 of 3 last visit is <0.2, and the difference between log HBsAg at 3 of 3 last visit and 1 of 3 last visit is <0.2.
Time Frame: Follow-up Week 48
Population: ITT population included participants who were randomly assigned or enrolled to an intervention arm and received at least 1 dose of intervention. Participants were analyzed according to study intervention they were randomly assigned or enrolled. Here "N" (Number of participants analyzed) signifies the number of participants that were evaluable for this OM.
Measure: Number; unit: Percentage of participants
Groups:
- FU Phase: Panel 1: After completion of OL phase (up to Week 48), Panel 1 participants enrolled prior to PA 5, entered FU phase and stopped JNJ-3989/JNJ-6379 and NA (if NA completion criteria [ALT <3*ULN, HBV DNA <LLOQ:20 IU/mL, HBeAg negative and HBsAg <10 IU/mL] was met as per Week 44 laboratory tests). If NA completion criteria were not met at OL Week 48, NA was continued till FU phase end (study Week 96). Participants on PegIN-alpha2a 180 mcg SC injection QW after Week 40 liver biopsy (for either 12 or 24 weeks) and who had not met NA completion criteria at Week 48 were assessed at PegIN-alpha2a treatment end and stopped NA, if NA completion criteria was met and then entered FU phase. If NA-retreatment criteria (HBV DNA >20,000 IU/mL, HBV DNA >2,000 IU/mL but <20,000 IU/mL & ALT >5*ULN) was met in FU phase, NA was re-started.
- FU Phase: Panel 2: After completion of OL phase (up to Week 48), Panel 2 participants enrolled prior to PA 5, entered FU phase and stopped JNJ-3989/JNJ-6379 and NA (if NA completion criteria [ALT <3*ULN, HBV DNA <LLOQ:20 IU/mL, HBeAg negative and HBsAg <10 IU/mL] was met as per Week 44 laboratory tests). If NA completion criteria were not met at OL Week 48, NA was continued till FU phase end (study Week 96). Participants on PegIN-alpha2a 180 mcg SC injection QW after Week 40 liver biopsy (for either 12 or 24 weeks) and who had not met NA completion criteria at Week 48 were assessed at PegIN-alpha2a treatment end and stopped NA, if NA completion criteria was met and then entered FU phase. If NA-retreatment criteria (HBV DNA >20,000 IU/mL, HBV DNA >2,000 IU/mL but <20,000 IU/mL & ALT >5*ULN) was met in FU phase, NA was re-started.
- FU Phase: Panel 3: After completion of OL phase (up to Week 48), Panel 3 participants enrolled per PA 5, entered FU phase and stopped JNJ-3989 and NA (if NA completion criteria [ALT <3*ULN, HBV DNA <LLOQ:20 IU/mL, HBeAg negative and HBsAg <10 IU/mL] was met as per Week 44 laboratory tests). If NA completion criteria were not met at OL Week 48, NA was continued till FU phase end (study Week 96). Participants on PegIN-alpha2a 180 mcg SC injection QW after Week 40 liver biopsy (for either 12 or 24 weeks) and who had not met NA completion criteria at Week 48 were assessed at PegIN-alpha2a treatment end and stopped NA, if NA completion criteria was met and then entered FU phase. If NA-retreatment criteria (HBV DNA >20,000 IU/mL, HBV DNA >2,000 IU/mL but <20,000 IU/mL & ALT >5*ULN) was met in FU phase, NA was re-started.
Arm/Group | FU Phase: Panel 1 | FU Phase: Panel 2 | FU Phase: Panel 3
Number analyzed (Participants) | 8 | 7 | 2
Percentage of participants | 50.0 [23.97 to 76.03] | 42.9 [16.96 to 72.14] | 50.0 [5.13 to 94.87]

9. Secondary Outcome: Panel 1, 2 and 3: Percentage of Participants Who Achieved HBsAg Seroclearance
Description: Percentage of Participants who achieved HBsAg Seroclearance were reported. HBsAg seroclearance was defined as quantitative HBsAg <LLOQ (<0.05 IU/mL).
Time Frame: Follow-up Week 48
Population: ITT population included participants who were randomly assigned or enrolled to an intervention arm and received at least 1 dose of intervention. Participants were analyzed according to study intervention they were randomly assigned or enrolled. Here "N" (Number of participants analyzed) signifies the number of participants that were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | FU Phase: Panel 1 | FU Phase: Panel 2 | FU Phase: Panel 3
Number analyzed (Participants) | 8 | 10 | 4
percentage of participants | 25.0 | 20.0 | 0

10. Secondary Outcome: Panel 1, 2 and 3: Percentage of Participants Who Achieved HBeAg Seroclearance
Description: Percentage of Participants who achieved HBeAg Seroclearance were reported. HBeAg seroclearance was defined as (quantitative] HBeAg <LLOQ (<0.11 IU/mL); with HBeAg positive status at baseline and became HBeAg negative post-baseline.
Time Frame: Follow-up Week 48
Population: ITT population: participants who were randomly assigned or enrolled to an intervention arm and received at least 1 dose of intervention. Participants were analyzed according to study intervention they were randomly assigned or enrolled. "N"(Number of participants analyzed) = number of participants evaluable for this outcome measure. Data was not collected for Panel 2 participants as they were HBeAg negative at enrollment and thus did not fulfill planned analysis criteria (HBeAg positive status).
Measure: Number; unit: percentage of participants
Arm/Group | FU Phase: Panel 1 | FU Phase: Panel 2 | FU Phase: Panel 3
Number analyzed (Participants) | 8 | 0 | 2
percentage of participants | 37.5 |  | 50.0

11. Secondary Outcome: Panel 1 and 2: Change From Baseline in Percentage of Intrahepatic Viral Parameter: Hepatitis B Core Antigen Positive (HBcAg+) Hepatocytes at Week 40
Description: Change from baseline in percentage of intrahepatic viral parameter: HBcAg positive hepatocytes at Week 40 were reported. The percentage of HBcAg positive hepatocytes were derived as number of HBcAg positive hepatocytes*100 per total number of evaluated hepatocytes.
Time Frame: Baseline, Week 40
Population: ITT population included participants who were randomly assigned or enrolled to an intervention arm and received at least 1 dose of intervention. Participants were analyzed according to study intervention they were randomly assigned or enrolled. Here "N" (Number of participants analyzed) signifies the number of participants that were evaluable for this outcome measure. Data for this OM was not planned to be collected and analyzed for Panel 3.
Measure: Median (Inter-Quartile Range); unit: percent change in HBcAg+ Hepatocytes
Arm/Group | Panel 1 | Panel 2
Number analyzed (Participants) | 6 | 9
percent change in HBcAg+ Hepatocytes | -54.49 [-87.02 to -42.26] | 0.03 [0.00 to 0.04]

12. Secondary Outcome: Panel 1,and 2: Change From Baseline in Percentage of Intrahepatic Viral Parameter: Covalently Closed Circular Deoxyribonucleic Acid Positive (cccDNA+) Hepatocytes at Week 40
Description: Change from baseline in percentage of intrahepatic viral parameter: cccDNA positive hepatocytes were reported. The percentage of cccDNA-positive hepatocytes, were derived as number of cccDNA positive hepatocytes*100 per total number of evaluated hepatocytes.
Time Frame: Baseline, Week 40
Population: ITT population included participants who were randomly assigned or enrolled to an intervention arm and received at least 1 dose of intervention. Participants were analyzed according to study intervention they were randomly assigned or enrolled. Here "N" (Number of participants analyzed) signifies the number of participants that were evaluable for this outcome measure. Data for this outcome measure was not planned to be collected and analyzed for Panel 3.
Measure: Median (Inter-Quartile Range); unit: percent change in cccDNA+ hepatocytes
Arm/Group | Panel 1 | Panel 2
Number analyzed (Participants) | 4 | 4
percent change in cccDNA+ hepatocytes | -4.50 [-40.88 to 12.97] | -2.40 [-22.84 to 7.57]

13. Secondary Outcome: Panel 1 and 2: Change From Baseline in Percentage of Intrahepatic Viral Parameter: HBsAg Positive (HBsAg+) Hepatocytes at Week 40
Description: Change from baseline in percentage of intrahepatic viral parameter: HBsAg positive hepatocytes at Week 40 were reported. The percentage of HBsAg positive hepatocytes were derived as number of HBsAg positive hepatocytes * 100 per total number of evaluated hepatocytes.
Time Frame: Baseline, Week 40
Population: ITT population included participants who were randomly assigned or enrolled to an intervention arm andreceived at least 1 dose of intervention. Participants were analyzed according to study intervention they were randomly assigned or enrolled. Here "N" (Number of participants analyzed) signifies the number of participants that were evaluable for this outcome measure. Data for this outcome measure was not planned to be collected and analyzed for Panel 3.
Measure: Median (Inter-Quartile Range); unit: percent change in HBsAg+ hepatocytes
Arm/Group | Panel 1 | Panel 2
Number analyzed (Participants) | 6 | 9
percent change in HBsAg+ hepatocytes | -92.38 [-95.65 to -73.37] | -14.19 [-21.11 to -7.01]

14. Secondary Outcome: Panel 1 and 2: Change From Baseline in Percentage of Intrahepatic Viral Parameter: Pre-genomic Ribonucleic Acid Positive (pgRNA+) Hepatocytes at Week 40
Description: Change from baseline in percentage of intrahepatic viral Parameter: pgRNA positive hepatocytes at Week 40 were reported. The percentage of pgRNA-positive hepatocytes, were derived as number of pgRNA positive hepatocytes*100 per total number of evaluated hepatocytes.
Time Frame: Baseline, Week 40
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: percent change in pgRNA+ hepatocytes
Arm/Group | Panel 1 | Panel 2
Number analyzed (Participants) | 4 | 4
percent change in pgRNA+ hepatocytes | -81.23 [-86.19 to -74.14] | -6.74 [-15.81 to -2.01]

15. Secondary Outcome: Panel 1 and 2: Change From Baseline in Transcriptional Activity (Ratio of pg RNA/cccDNA) at Week 40
Description: Change from baseline in transcriptional activity (ratio of pgRNA/cccDNA) at Week 40 were reported.
Time Frame: Baseline, Week 40
Population: as for outcome 12
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Panel 1 | Panel 2
Number analyzed (Participants) | 4 | 4
ratio | 50.00 [49.07 to 58.83] | 8.86 [-3.03 to 27.45]

16. Secondary Outcome: Panel 1, 2: Change From Baseline in Percentage of Intrahepatic Viral Parameter: Silent Infected Hepatocytes at Week 40
Description: Change from baseline in percentage of intrahepatic viral parameter: silent infected hepatocytes (that is infected hepatocytes without HBV transcription; cccDNA-positive/HBV RNA-negative hepatocytes) at Week 40 were reported. The percentage of silent infected hepatocytes (SIH), were derived as number of silent infected hepatocytes*100 per total number of evaluated hepatocytes.
Time Frame: Baseline, Week 40
Population: as for outcome 12
Measure: Median (Inter-Quartile Range); unit: percent change in SIH
Arm/Group | Panel 1 | Panel 2
Number analyzed (Participants) | 4 | 4
percent change in SIH | 25.06 [21.40 to 31.63] | 2.88 [-14.74 to 8.80]

17. Secondary Outcome: Panel 1, 2 and 3: Percentage of Participants With HBsAg Seroclearance at Week 72 Without Restarting Nucleos(t)Ide Analog (NA) Treatment
Description: Percentage of participants with HBsAg seroclearance (defined as HBsAg < LLOQ: 0.05 IU/mL) at Week 72 without restarting NA treatment were reported.
Time Frame: At Week 72 (24 weeks after completion of all study drugs at Week 48)
Population: ITT population included participants who were randomly assigned or enrolled to an intervention arm and received at least 1 dose of intervention. Participants were analyzed according to study intervention they were randomly assigned or enrolled. Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Groups:
- FU Phase: Panel 1: After completion of OL phase (up to Week 48) all Panel 1 participants enrolled prior to PA 5, entered FU phase and stopped JNJ-3989/JNJ-6379 and NA (if NA completion criteria [ALT <3*ULN, HBV DNA <LLOQ:20 IU/mL, HBeAg negative and HBsAg <10 IU/mL] was met as per Week 44 laboratory tests). If NA completion criteria were not met at OL Week 48, NA was continued till FU phase end (study Week 96). Participants on PegIN-alpha2a 180 mcg SC injection QW after Week 40 liver biopsy (for either 12 or 24 weeks) and who had not met NA completion criteria at Week 48 were assessed at PegIN-alpha2a treatment end and stopped NA, if NA completion criteria was met and then entered FU phase. If NA-retreatment criteria (HBV DNA >20,000 IU/mL, HBV DNA >2,000 IU/mL but <20,000 IU/mL & ALT >5*ULN) was met in FU phase, NA was re-started.
Arm/Group | FU Phase: Panel 1 | FU Phase: Panel 2 | FU Phase: Panel 3
Number analyzed (Participants) | 9 | 10 | 4
Percentage of participants | 0 | 1 | 0

18. Secondary Outcome: Panel 1, 2 and 3: Percentage of Participants With Sustained (Reduction) Serum HBsAg Response Per Definition 1 at Follow-up Week 48
Description: Percentage of participants with sustained (reduction) serum HBsAg response per Definition 1 at follow-up Week 48 were reported. Sustained serum HBsAg response per definition 1 was defined as: for participants with data for last follow-up visit (Follow-up Week 48 for participants who did not receive PegIFN-alpha2a or received PegIFN-alpha2a and did not meet NA completion criteria, and last Follow-up visit for participants who received PegIFN-alpha2a and stopped NA during Follow-up): participants who had a >1 log decline in HBsAg response at last scheduled follow-up visit and had an HBsAg <1000 IU/mL at last scheduled follow-up visit, or for participants without data at last follow-up visit: HBsAg values had a >2 log decline at second most recent visit or >1.5 log decline at latest visit (most recent value used) compared to baseline and had an HBsAg <1000 IU/mL at last available timepoint.
Time Frame: Follow-up Week 48
Population: ITT population included participants who were randomly assigned or enrolled to an intervention arm and received at least 1 dose of intervention. Participants were analyzed according to study intervention they were randomly assigned or enrolled.
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | FU Phase: Panel 1 | FU Phase: Panel 2 | FU Phase: Panel 3
Number analyzed (Participants) | 10 | 10 | 4
Percentage of participants | 50.0 [26.73 to 73.27] | 70.0 [44.83 to 88.42] | 50.0 [14.26 to 85.74]

19. Secondary Outcome: Panel 1, 2 and 3: Percentage of Participants With Sustained (Reduction) Serum HBsAg Response Per Definition 3 at Follow-up Week 48
Description: Percentage of participants with sustained (reduction) serum HBsAg response per Definition 3 at follow-up Week 48 were reported. Sustained serum HBsAg response per definition 3 for participants with a >1 log decline in HBsAg from baseline at last follow up visit: Among the most recent three visits, the difference between log HBsAg at 2 of 3 last visit and 1 of 3 last visit is <0.2, and the difference between log HBsAg at 3 of 3 last visit and 1 of 3 last visit is <0.2 and have an HBsAg <1000 IU/mL at the last available timepoint.
Time Frame: From follow-up Week 24 up to follow-up Week 48
Population: as for outcome 9
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | FU Phase: Panel 1 | FU Phase: Panel 2 | FU Phase: Panel 3
Number analyzed (Participants) | 8 | 7 | 2
Percentage of participants | 25.0 [6.86 to 53.82] | 42.9 [16.96 to 72.14] | 50.0 [5.13 to 94.87]

20. Secondary Outcome: Panel 1, 2 and 3: Percentage of Participants With Sustained (Reduction) Serum HBsAg Response Per Definition 4 at Follow-up Week 48
Description: Percentage of participants with sustained (reduction) serum HBsAg response per definition 4 follow-up Week 48 were reported. Sustained serum HBsAg response per definition 4 were classified into 3 categories with respect to the difference between HBsAg level at the last Follow-up timepoint and end of treatment: Increase: >+0.2 log10 IU/mL , stable: within plus or minus (+/-) 0.2 log10 IU/mL, and decrease: >-0.2 log10 IU/mL.
Time Frame: Follow-up Week 48
Population: as for outcome 9
Measure: Number; unit: Percentage of participants
Arm/Group | FU Phase: Panel 1 | FU Phase: Panel 2 | FU Phase: Panel 3
Number analyzed (Participants) | 9 | 10 | 4
Percentage of participants
  Stable: Within +/-0.2 log10 | 11.1 | 0 | 0
  Decrease: > -0.2 log10 IU/mL | 22.2 | 30.0 | 25.0
  Increase: > +0.2 log10 IU/mL | 66.7 | 70.0 | 75.0

21. Secondary Outcome: Panel 1, 2 and 3: Percentage of Participants Who Achieved HBsAg Seroconversion
Description: Seroconversion of HBsAg was defined as having achieved HBsAg seroclearance (defined as quantitative HBsAg <LLOQ [<0.05 IU/mL]) and appearance of anti-HBs antibodies (defined as a baseline anti-HBs antibodies [quantitative] <LLOQ [<5 milli-international units per milliliter {mIU/mL}] and a post-baseline assessment >=LLOQ [>=5 mIU/mL]).
Time Frame: From baseline (Day 1) up to follow-up Week 48
Population: as for outcome 17
Measure: Number; unit: Percentage of participants
Arm/Group | Panel 1 | Panel 2 | Panel 3
Number analyzed (Participants) | 7 | 9 | 4
Percentage of participants | 28.6 | 11.1 | 0

22. Secondary Outcome: Panel 1, 2 and 3: Percentage of Participants Who Achieved HBeAg Seroconversion
Description: Percentage of participants who achieved HBeAg seroconversion were reported. Seroconversion of HBeAg was defined as having achieved HBeAg seroclearance (defined as [quantitative] HBeAg <LLOQ [<0.11 IU/mL]; with HBeAg positive status at baseline and became HBeAg negative post-baseline) together with appearance of anti-HBe antibodies (defined as a baseline anti-HBe antibodies [qualitative] with a "negative" result and a post-baseline assessment with "positive" result).
Time Frame: From baseline (Day 1) up to follow-up Week 48
Population: ITT population: participants randomly assigned or enrolled to an intervention arm and received at least 1 dose of intervention. Participants were analyzed according to study intervention they were randomly assigned or enrolled. "N' (number of participants analyzed) = participants evaluable for this outcome measure. Data was not collected for Panel 2 participants as they were HBeAg negative at enrollment and thus did not fulfill planned analysis criteria (HBeAg positive status).
Measure: Number; unit: Percentage of participants
Arm/Group | Panel 1 | Panel 2 | Panel 3
Number analyzed (Participants) | 7 | 0 | 2
Percentage of participants | 28.6 |  | 50.0

23. Secondary Outcome: Panel 1, 2 and 3: Percentage of Participants With Off-treatment Virologic Flares Per Derivation 1
Description: Virologic flare (VF) per derivation 1 was defined only for participants who were off-treatment (period after stopping all study drugs, including NA) and who had HBV DNA<LLOQ (<20 IU/mL) at last observed point on-treatment [OT]); start date of confirmed VF was first date of 2 consecutive visits with HBV DNA >200 IU/mL. End date of same confirmed VF was first date when HBV DNA value returns to <=200 IU/mL or date of NA restart, whichever comes first. Each virologic flare were categorized based on confirmed (that is, 2 consecutive values) peak HBV DNA above any of 3 thresholds within the start and end date of that flare as followed: 20,000 IU/mL, 2,000 IU/mL, and 200 IU/mL. Participants were counted only once for any given flare, regardless of the number of times they actually experienced the flare.
Time Frame: From baseline (Day 1) up to follow-up Week 48
Population: ITT population: participants randomly assigned or enrolled to an intervention arm and received at least 1 dose of drug. Participants were analyzed according to study drug randomly assigned/enrolled. "N" (Number of participants analyzed) = participants evaluable for this outcome measure. Data was not collected for Panel 1, as no participants met off-treatment criteria (set duration between last dose and last study visit) at final analysis and thus were not considered eligible for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Panel 1 | Panel 2 | Panel 3
Number analyzed (Participants) | 0 | 3 | 2
percentage of participants
  HBV DNA > 200 IU/mL |  | 0 | 0
  HBV DNA > 2,000 IU/mL |  | 33.3 | 0
  HBV DNA > 20,000 IU/mL |  | 0 | 50.0

24. Secondary Outcome: Panel 1, 2 and 3: Percentage of Participants With Off-treatment and On-treatment Biochemical Flares
Description: Off-treatment (time period after stopping all study drugs [including NA]) biochemical flare was defined as first date of 2 consecutive visits with ALT and/or AST >=3*ULN and >=3*nadir (lowest value observed up to start of flare) while participant received no study drugs. End date of same off-treatment biochemical flare was defined as first date with 50 percentage (%) reduction from peak ALT and/or AST level & <3*ULN. On-treatment (time period during which the participant received any of study drugs) biochemical flare was defined as first date of 2 consecutive visits with ALT and/or AST >=3*ULN and >=3*nadir (lowest value observed up to start of flare) while participant was on-treatment. End date of same on-treatment biochemical flare was defined as first date with a 50% reduction from the peak ALT and/or AST level and <3*ULN, regardless of stopping study drugs. Participants were counted only once for any given flare, regardless of the number of times they actually experienced flare.
Time Frame: From baseline (Day 1) up to follow-up Week 48
Population: ITT population included participants who were randomly assigned or enrolled to an intervention arm and received at least 1 dose of intervention. Participants were analyzed according to study intervention they were randomly assigned or enrolled. Here, "n"(number analyzed) signifies number of participants analyzed at specified categories and n=0 signifies that no participant was available for the analysis at the specified category.
Measure: Number; unit: percentage of participants
Arm/Group | Panel 1 | Panel 2 | Panel 3
Number analyzed (Participants) | 10 | 10 | 4
percentage of participants
  Off-treatment biochemical flare: number analyzed (Participants) | 0 | 3 | 2
  Off-treatment biochemical flare |  | 0 | 0
  On-treatment biochemical flare | 10.0 | 10.0 | 25.0

25. Secondary Outcome: Panel 1, 2 and 3: Percentage of Participants With Off-treatment Clinical Flares
Description: Percentage of participants with off-treatment clinical flares were reported. Clinical flares occurred either when a virologic flare and biochemical flare overlapped in time or when a biochemical flare started within 4 weeks following the end of a virologic flare. Off-treatment was defined as the time period after stopping all study drugs (including NA). The start date of a clinical flare was the minimum start date of the virologic flare and biochemical flare. The end date of a clinical flare was the maximum end date of the virologic flare and biochemical flare, that is, the later date between HBV DNA returned to <=200 IU/mL (or <=1 log10) and 50 %reduction from the peak ALT and/or AST level and <3*ULN reached during the biochemical flare. Participants were counted only once for any given flare, regardless of the number of times they actually experienced the flare.
Time Frame: From baseline (Day 1) up to follow-up Week 48
Population: ITT population: participants randomly assigned/enrolled to an intervention arm and received at least 1 dose of drug. Participants were analyzed according to study drug randomly assigned/enrolled. "N" (Number of participants analyzed) = participants evaluable for this outcome measure. Data was not collected for Panel 1, as no participants met off-treatment criteria (set duration between last dose and last study visit) at final analysis and thus were not considered eligible for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Panel 1 | Panel 2 | Panel 3
Number analyzed (Participants) | 0 | 3 | 2
percentage of participants
  HBV DNA >200 IU/mL |  | 0 | 0
  HBV DNA >2,000 IU/mL |  | 0 | 0
  HBV DNA >20,000 IU/mL |  | 0 | 50.0

26. Secondary Outcome: Panel 1, 2 and 3: Time to First Occurence of HBsAg Seroclearance
Description: Time to first occurrence of HBsAg seroclearance (defined as quantitative HBsAg <LLOQ [<0.05 IU/mL]) were reported. Time to first occurrence of HBsAg seroclearance was defined as the number of days between the date of first study intervention intake and the date of the first occurrence of the HBsAg seroclearance. Participants who withdrew early from the study before achieving HBsAg seroclearance or who did not achieve HBsAg seroclearance were censored at the last available HBsAg assessment. Kaplan-Meier method was used for the estimation.
Time Frame: From baseline (Day 1) up to follow-up Week 48
Population: as for outcome 18
Measure: Median (80% Confidence Interval); unit: weeks
Arm/Group | Panel 1 | Panel 2 | Panel 3
Number analyzed (Participants) | 10 | 10 | 4
weeks | NA [NA to NA] — NA indicates that median and 80% CI data were not estimable due to insufficient number of participants with events. | NA [NA to NA] — NA indicates that median and 80% CI data were not estimable due to insufficient number of participants with events. | NA [NA to NA] — NA indicates that median and 80% CI data were not estimable due to insufficient number of participants with events.

27. Secondary Outcome: Panel 1, 2 and 3: Percentage of Participants With Virologic Breakthrough
Description: Percentage of participants with virologic breakthrough on treatment were reported. Virological breakthrough was defined as having a confirmed on-treatment HBV DNA increase by >1 log10 IU/mL from nadir level (lowest level reached during treatment) in participants who did not have on-treatment HBV DNA level < LLOQ (<20 IU/mL) or confirmed on-treatment HBV DNA level >200 IU/mL in participants who had on-treatment HBV DNA level <LLOQ (<20 IU/mL) of the HBV DNA assay. Confirmed HBV DNA increase/level means that the criterion should be fulfilled at 2 or more consecutive time points or at the last observed on-treatment time point. On treatment was defined as the time period in which the participant received any of the study interventions (JNJ-3989 and/or JNJ 6379 and/or NA and/or PegIFN-alpha2a).
Time Frame: From baseline (Day 1) up to follow-up Week 48
Population: as for outcome 18
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Panel 1 | Panel 2 | Panel 3
Number analyzed (Participants) | 10 | 10 | 4
percentage of participants | 0 [0.00 to 20.57] | 0 [0.00 to 20.57] | 0 [0.00 to 43.77]

28. Secondary Outcome: Panel 1, 2 and 3: Percentage of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: Percentage of participants with TEAES (including serious and non-serious) and TESAEs were reported. An AE was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. Any AE occurring at or after the initial administration of study intervention was considered to be treatment emergent. A SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Open-label: Day 1 (Week 1) up to Week 48; Follow-up Phase: Follow-up Week 1 up to follow-up Week 48
Population: Safety analysis set included all participants who received at least 1 dose of study intervention. Participants were analyzed according to the study intervention they actually received.
Measure: Number; unit: percentage of participants
Groups:
- OL Phase: Panel 1: Prior to PA 5, participants received either JNJ-3989 200 mg SC injection Q4W from Day 1 (Week 1) to Week 44 + JNJ-6379 250 mg QD + NA (ETV 0.5 mg/TD 245 mg/TAF 25 mg) QD from Day 1 (Week 1) to Week 48 or JNJ-3989 200 mg SC injection Q4W from Day 1 (Week 1) to Week 44+NA (ETV 0.5 mg/TD 245 mg/TAF 25 mg) QD from Day 1 (Week 1) to Week 48. After PA 5, participants stopped JNJ-6379 and continued JNJ-3989+NA. With separate consent, participants received optional treatment: PegIFN-alpha-2a 180 mcg SC injection QW post Week 40 liver biopsy for either 12 or 24 weeks (anytime between study Week 40 to 72) at investigator's discretion. At end of treatment Week 48, all participants entered FU phase and stopped JNJ-3989/JNJ-6379 and NA (if NA completion criteria [ALT <3*ULN, HBV DNA <LLOQ:20 IU/mL, HBeAg negative and HBsAg <10 IU/mL] was met as per Week 44 laboratory tests). If NA completion criteria were not met at Week 48, NA was continued till FU phase end (study Week 96).
- OL Phase: Panel 2: Prior to PA 5, participants received either JNJ-3989 200 mg SC injection Q4W from Day 1 (Week 1) to Week 44 + JNJ-6379 250 mg QD and NA treatment (ETV 0.5 mg/TD 245 mg/TAF 25 mg) QD from Day 1 (Week 1) to Week 48, or JNJ-3989 200 mg SC injection Q4W from Day 1 (Week 1) to Week 44 + NA (ETV 0.5 mg/TD 245 mg/TAF 25 mg) QD from Day 1 (Week 1) to Week 48. After PA 5, participants discontinued JNJ-6379 and continued JNJ-3989 + NA. With separate consent, participants received optional treatment with PegIFN-alpha-2a 180 mcg SC injection QW after Week 40 liver biopsy for either 12 or 24 weeks (anytime between study Week 40 to 72) at investigator's discretion. At end of treatment Week 48, all participants entered FU phase and stopped JNJ-3989/JNJ-6379 and NA (if NA treatment completion criteria [ALT <3*ULN, HBV DNA <LLOQ; 20 IU/mL, HBeAg negative and HBsAg <10 IU/mL] was met as per Week 44 laboratory tests). If NA completion criteria were not met at Week 48, NA was continued till FU phase end (study Week 96).
- OL Phase: Panel 3: After PA 5, participants received either JNJ-3989 200 mg SC injection Q4W from Day 1 (Week 1 to Week 44) + JNJ-6379 250 mg QD and NA treatment (ETV 0.5 mg/TD 245 mg/TAF 25 mg) QD from Day 1 (Week 1) to Week 48, or JNJ-3989 200 mg SC injection Q4W from Day 1 (Week 1) to Week 44 + NA (ETV 0.5 mg/TD 245 mg/TAF 25 mg) QD from Day 1 (Week 1) to Week 48. After PA 5, participants discontinued JNJ-6379 and continued JNJ-3989 + NA. With separate consent, participants received optional treatment with PegIFN-alpha-2a 180 mcg SC injection QW after Week 40 liver biopsy for either 12 or 24 weeks (anytime between study Week 40 to 72) at investigator's discretion. At end of treatment Week 48, all participants entered FU phase and stopped JNJ-3989/JNJ-6379 and NA (if NA treatment completion criteria [ALT <3*ULN, HBV DNA <LLOQ; 20 IU/mL, HBeAg negative and HBsAg <10 IU/mL] was met as per Week 44 laboratory tests). If NA completion criteria were not met at Week 48, NA was continued till FU phase end (study Week 96).
Arm/Group | OL Phase: Panel 1 | OL Phase: Panel 2 | OL Phase: Panel 3 | FU Phase: Panel 1 | FU Phase: Panel 2 | FU Phase: Panel 3
Number analyzed (Participants) | 10 | 10 | 4 | 10 | 10 | 4
percentage of participants
  TEAEs | 90.0 | 100.0 | 75.0 | 50.0 | 60.0 | 75.0
  TESAEs | 10.0 | 0 | 0 | 0 | 0 | 0

29. Secondary Outcome: Panel 1, 2 and 3: Number of Participants With HBV-Specific Peripheral Blood T-cell Responses
Description: Number of participants with HBV-specific peripheral blood T-cell responses were reported. HBV-specific T-cells were characterized in peripheral blood mononuclear cell immune analysis by binding assays (multimer staining) combined with downstream T-cell responses and transcriptome profiling.
Time Frame: Open-label: Weeks 40, 44, and 48; Follow-up Phase: Follow-up Weeks 2, 12 and 24
Population: ITT population were analyzed. Participants were analyzed according to study intervention they were randomly assigned or enrolled. Here "N" (Number of participants analyzed) signifies the number of participants that were evaluable for this outcome measure and "n"(number analyzed) signifies number of participants analyzed at specified categories. Here, n=0, signifies that no participants were available for the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | OL Phase: Panel 1 | OL Phase: Panel 2 | OL Phase: Panel 3 | FU Phase: Panel 1 | FU Phase: Panel 2 | FU Phase: Panel 3
Number analyzed (Participants) | 7 | 7 | 1 | 9 | 10 | 4
Participants
  Open Label: Week 40: number analyzed (Participants) | 7 | 7 | 1 | 0 | 0 | 0
  Open Label: Week 40 | 6 | 6 | 0 |  |  |
  Open Label: Week 44: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0 | 0
  Open Label: Week 44 | 0 | 1 |  |  |  |
  Open Label: Week 48: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  Open Label: Week 48 | 1 |  |  |  |  |
  Follow-up Week 2: number analyzed (Participants) | 0 | 0 | 0 | 8 | 10 | 3
  Follow-up Week 2 |  |  |  | 4 | 10 | 3
  Follow-up Week 12: number analyzed (Participants) | 0 | 0 | 0 | 3 | 7 | 3
  Follow-up Week 12 |  |  |  | 1 | 5 | 2
  Follow-up Week 24: number analyzed (Participants) | 0 | 0 | 0 | 9 | 9 | 4
  Follow-up Week 24 |  |  |  | 5 | 9 | 4

30. Secondary Outcome: Panel 1, 2 and 3: Percentage of Participants With Worst (Grade 3 and 4) Treatment-emergent Division of Acquired Immunodeficiency Syndrome (DAIDS) Toxicity Grade in Clinical Laboratory Tests
Description: Clinical laboratory test parameters were Hematology : absolute neutrophil count (ANC); Chemistry : alanine aminotransferase (ALT) and serum glutamic pyruvic transaminase (SGPT), aspartate aminotransferase(AST) or serum glutamic oxaloacetic transaminase (SGOT), amylase (pancreatic and total), creatinine Kinase, creatinine, low-density lipoprotein (LDL), lipase, estimated glomerular filtration rate (eGFR) on serum creatinine (Cr). DAIDS toxicity grades were Grade 1 (Mild), Grade 2 (Moderate), Grade 3 (Severe), Grade 4 (Potentially Life-Threatening). Percentage of participants with treatment-emergent DAIDS toxicity Grade 3 or 4 were reported in this outcome measure. For toxicity grades, treatment-emergent was concluded if the postbaseline grade was worse than the baseline grade. Only those abnormality categories in which at least one participant had data were reported.
Time Frame: Open-label: Day 1 (Week 1) up to Week 48; Follow-up Phase: Follow-up Week 1 up to follow-up Week 48
Population: Safety analysis set included all participants who received at least 1 dose of study intervention. Participants were analyzed according to the study intervention they actually received. Here "n" (number analyzed) signifies number of participants analyzed at specified categories.
Measure: Number; unit: percentage of participants
Arm/Group | OL Phase: Panel 1 | OL Phase: Panel 2 | OL Phase: Panel 3 | FU Phase: Panel 1 | FU Phase: Panel 2 | FU Phase: Panel 3
Number analyzed (Participants) | 10 | 10 | 4 | 10 | 10 | 4
percentage of participants
  Hematology: Absolute Neutrophil Count: Low: Grade 3: number analyzed (Participants) | 9 | 10 | 4 | 10 | 10 | 4
  Hematology: Absolute Neutrophil Count: Low: Grade 3 | 0 | 10.0 | 25.0 | 0 | 10.0 | 25.0
  Chemistry: ALT or SGPT: High: Grade 3: number analyzed (Participants) | 9 | 10 | 4 | 10 | 10 | 4
  Chemistry: ALT or SGPT: High: Grade 3 | 0 | 10.0 | 25.0 | 10.0 | 10.0 | 0
  Chemistry: ALT or SGPT: High: Grade 4: number analyzed (Participants) | 9 | 10 | 4 | 10 | 10 | 4
  Chemistry: ALT or SGPT: High: Grade 4 | 0 | 0 | 0 | 0 | 0 | 25.0
  Chemistry: AST/SGOT: High: Grade 3: number analyzed (Participants) | 9 | 10 | 4 | 10 | 10 | 4
  Chemistry: AST/SGOT: High: Grade 3 | 0 | 10.0 | 0 | 0 | 0 | 25.0
  Chemistry: Amylase (Pancreatic): High: Grade 4: number analyzed (Participants) | 4 | 5 | 4 | 4 | 5 | 3
  Chemistry: Amylase (Pancreatic): High: Grade 4 | 25.0 | 0 | 0 | 0 | 0 | 0
  Chemistry: Amylase (Total): High: Grade 3: number analyzed (Participants) | 9 | 10 | 4 | 9 | 10 | 4
  Chemistry: Amylase (Total): High: Grade 3 | 11.1 | 0 | 0 | 0 | 0 | 0
  Chemistry: Creatinine Kinase : High: Grade 3: number analyzed (Participants) | 9 | 10 | 4 | 10 | 10 | 4
  Chemistry: Creatinine Kinase : High: Grade 3 | 0 | 0 | 25.0 | 0 | 0 | 0
  Chemistry: Creatinine Kinase : High: Grade 4: number analyzed (Participants) | 9 | 10 | 4 | 10 | 10 | 4
  Chemistry: Creatinine Kinase : High: Grade 4 | 0 | 10.0 | 0 | 0 | 0 | 0
  Chemistry: Creatinine: High: Grade 3: number analyzed (Participants) | 9 | 10 | 4 | 10 | 10 | 4
  Chemistry: Creatinine: High: Grade 3 | 11.1 | 0 | 0 | 0 | 0 | 0
  Chemistry: LDL (Fasting): High: Grade 3: number analyzed (Participants) | 9 | 10 | 4 | 9 | 10 | 4
  Chemistry: LDL (Fasting): High: Grade 3 | 0 | 10.0 | 0 | 0 | 0 | 0
  Chemistry: Lipase: High: Grade 3: number analyzed (Participants) | 9 | 10 | 4 | 9 | 10 | 4
  Chemistry: Lipase: High: Grade 3 | 0 | 10.0 | 0 | 0 | 0 | 0
  Chemistry: eGFR Cr: Low: Grade 3: number analyzed (Participants) | 9 | 10 | 4 | 10 | 10 | 4
  Chemistry: eGFR Cr: Low: Grade 3 | 0 | 10.0 | 0 | 0 | 0 | 0

31. Secondary Outcome: Panel 1, 2 and 3: Percentage of Participants With Worst (Abnormally Low/High)Treatment-emergent DAIDS Toxicity Grade in Electrocardiogram (ECG)
Description: ECG parameters included ECG mean heart rate (HR)(beats per minute[bpm]), Pulse rate (PR) interval (milliseconds [ms]), QRS duration (ms) and QTc Corrected (Fridericia's formula QTcF). Abnormalities were graded as follows: ECG mean heart rate (abnormally low HR <45 bpm) and (abnormally high HR>=120 bpm); PR interval (abnormally high >220 ms) and QPRS (abnormally high >=120 ms); OT interval corrected for heart rate according to Fridericia (QTcF); borderline prolonged (BRD Pr )QTc (>=450 to <=480 ms), prolonged QTc (>=480 to <=500 ms)and pathologically prolonged QTc (>500 ms). For worst abnormality, treatment-emergent was concluded if the abnormality worsened as compared to the abnormality at baseline: abnormally high to abnormally low and vice-versa. Only those abnormality categories in which at least one participant had data were reported.
Time Frame: Open-label: Day 1 (Week 1) up to Week 48; Follow-up Phase: Follow-up Week 1 up to follow-up Week 48
Population: Safety analysis set included all participants who received at least 1 dose of study intervention. Participants were analyzed according to the study intervention they actually received. Here "N" (Number of participants analyzed) signifies the number of participants that were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | OL Phase: Panel 1 | OL Phase: Panel 2 | OL Phase: Panel 3 | FU Phase: Panel 1 | FU Phase: Panel 2 | FU Phase: Panel 3
Number analyzed (Participants) | 9 | 10 | 4 | 9 | 10 | 4
percentage of participants
  ECG Mean HR: low (<45 bpm) | 0 | 10.0 | 0 | 0 | 10.0 | 0
  PR Interval: Aggregate: Abnormally high (>220 ms) | 11.1 | 20.0 | 0 | 11.1 | 20.0 | 0
  QTcF Interval: Aggregate: borderline prolonged QT (>=450to<=480 ms) | 0 | 10.0 | 0 | 0 | 0 | 0

32. Secondary Outcome: Panel 1, 2 and 3: Percentage of Participants With Worst (Abnormally Low/High) Treatment-emergent DAIDS Toxicity Grade in Vital Signs
Description: Percentage of participants with worst treatment-emergent DAIDS toxicity grade in vital signs were reported. Abnormality grades were: pulse rate (abnormally low <=45 bpm) and (abnormally high >=120 bpm). An assessment was treatment-emergent if abnormality worsened as compared to the abnormality at baseline: from abnormally high to abnormally low and vice-versa. Only the category (pulse rate) in which at least one participant had data were reported.
Time Frame: Open-label: Day 1 (Week 1) up to Week 48; Follow-up Phase: Follow-up Week 1 up to follow-up Week 48
Population: Safety analysis set included all participants who received at least 1 dose of study intervention. Participants were analyzed according to the study intervention they actually received. Here "N" (Number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | OL Phase: Panel 1 | OL Phase: Panel 2 | OL Phase: Panel 3 | FU Phase: Panel 1 | FU Phase: Panel 2 | FU Phase: Panel 3
Number analyzed (Participants) | 9 | 10 | 4 | 10 | 10 | 4
percentage of participants | 0 | 10.0 | 0 | 0 | 0 | 0

33. Secondary Outcome: Panel 1, 2 and 3: Number of Participants With Clinically Significant Treatment-emergent Abnormalities in Physical Examination
Description: Number of participants with clinically significant treatment-emergent abnormalities in physical examination were reported. Physical examination included head/neck/thyroid, eyes/ears/nose/throat, respiratory, cardiovascular, lymph nodes, abdomen, skin, musculoskeletal, and neurological examinations.
Time Frame: Open-label: Day 1 (Week 1) up to Week 48; Follow-up Phase: Follow-up Week 1 up to follow-up Week 48
Population: as for outcome 28
Measure: Count of Participants; unit: Participants
Arm/Group | OL Phase: Panel 1 | OL Phase: Panel 2 | OL Phase: Panel 3 | FU Phase: Panel 1 | FU Phase: Panel 2 | FU Phase: Panel 3
Number analyzed (Participants) | 10 | 10 | 4 | 10 | 10 | 4
Participants | 4 | 0 | 0 | 0 | 0 | 0

34. Secondary Outcome: Panel 2 and 3: Plasma Trough Concentration (C[0hour]) of JNJ-73763989 (JNJ-73763976, JNJ-73763924)
Description: Plasma trough concentration (C[0hour]) of JNJ-73763989 (JNJ-73763976, JNJ-73763924) were reported. C0h was the pre-dose plasma concentration of the JNJ-73763989 (JNJ-73763976, JNJ-73763924). Non-compartmental analysis were conducted to analyze plasma concentration of JNJ-73763989 and its molecules.
Time Frame: Week 4 : Pre-dose on Day 29
Population: A pharmacokinetics (PK) analysis which included participants of Panel 2 and Panel 3 who had consented to participate in the intensive PK subgroup were analyzed. Data for this outcome measure was planned to be collected and analyzed for Panel 2 and 3 alone.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Panel 2 | Panel 3
Number analyzed (Participants) | 3 | 4
nanograms per milliliter (ng/mL)
  JNJ-73763976 | NA (NA) — NA signifies that mean and standard deviation were not calculable because sample concentration was below quantification limit (that is <2.1 ng/mL). | NA (NA) — NA signifies that mean and standard deviation were not calculable because sample concentration was below quantification limit (that is <2.1 ng/mL).
  JNJ-73763924 | NA (NA) — NA signifies that mean and standard deviation were not calculable because sample concentration was below quantification limit (that is <2.1 ng/mL). | NA (NA) — NA signifies that mean and standard deviation were not calculable because sample concentration was below quantification limit (that is <2.1 ng/mL).

35. Secondary Outcome: Panel 2: Maximum Observed Plasma Concentration (Cmax) of JNJ-73763989 (JNJ-73763976, JNJ-73763924)
Description: Maximum observed plasma concentration (Cmax) of JNJ-73763989 (JNJ-73763976, JNJ-73763924) were reported. Non-compartmental analysis were conducted to analyze Cmax JNJ-73763989 and its molecules.
Time Frame: Week 4 (Day 29): Pre-dose and 15 minutes, 30 minutes, 1, 2, 3, 4, 6, 8, 10 and 24 hours post dose
Population: Pharmacokinetics (PK) analysis included Panel 2 participants who had consented to participate in intensive PK subgroup. "N" (Number of participants analyzed) = participants who were evaluable for this outcome measure. "n"(number analyzed) = number of participants analyzed at specified categories. As planned, summary analysis was performed when overall number of participants analyzed were >=3 and thus participant wise data were reported for Panel 2 alone in this outcome measure.
Measure: Number; unit: nanograms per milliliter (ng/mL)
Groups:
- Panel 2: Prior to PA 5, participants received either JNJ-3989 200 mg SC injection Q4W from Day 1 (Week] 0 to Week 44 + JNJ-6379 250 mg tablet QD and NA treatment (ETV 0.5 mg, TD 245 mg/TAF 25 mg) tablet QD from Day 1 (Week 0) to Week 48, or JNJ-3989 200 mg SC injection Q4W (from Day 1 [Week 0] to Week 44) + NA (ETV 0.5 mg/TD 245 mg/TAF 25 mg) tablet QD from Day 1 (Week 0) to Week 48. After PA 5, participants discontinued JNJ-6379 but continued treatment with JNJ-3989 + NA (ETV, TD, or TAF). Participants with a separate consent started optional treatment with PegIFN-alpha-2a 180 mcg SC injection QW started after Week 40 liver biopsy for 12 or 24 weeks (till study Week 60 or 72) at investigator's discretion. At Week 48, all participants entered follow-up and stopped all study drugs, but NA was continued till end of follow-up (study Week 96) if NA treatment completion criteria (ALT <3*ULN, HBV DNA <LLOQ; 20 IU/mL, HBeAg negative and HBsAg <10 IU/mL) was not met at Week 48. Participants who met NA treatment completion criteria (at Week 48) were monitored Q4W in the follow-up phase. If NA-retreatment criteria (HBV DNA >20,000 IU/mL, HBV DNA >2,000 IU/mL but <20,000 IU/mL & ALT >5*ULN) was met, NA retreatment was started.
Arm/Group | Panel 2
Number analyzed (Participants) | 2
nanograms per milliliter (ng/mL)
  JNJ-73763976 - Participant 1: number analyzed (Participants) | 1
  JNJ-73763976 - Participant 1 | 2757
  JNJ-73763976 - Participant 2: number analyzed (Participants) | 1
  JNJ-73763976 - Participant 2 | 1062
  JNJ-73763924 - Participant 1: number analyzed (Participants) | 1
  JNJ-73763924 - Participant 1 | 595
  JNJ-73763924 - Participant 2: number analyzed (Participants) | 1
  JNJ-73763924 - Participant 2 | 205

36. Secondary Outcome: Panel 3: Maximum Observed Plasma Concentration (Cmax) of JNJ-73763989 (JNJ-73763976, JNJ-73763924)
Description: as for outcome 35
Time Frame: Week 4 (Day 29): Pre-dose and 15 minutes, 30 minutes, 1, 2, 3, 4, 6, 8, 10 and 24 hours post dose
Population: Pharmacokinetics (PK) analysis which included Panel 3 participants who had consented to participate in the intensive PK subgroup. Data for this outcome measure was planned to be collected and analyzed for Panel 3 alone.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Panel 3
Number analyzed (Participants) | 4
nanograms per milliliter (ng/mL)
  JNJ-73763976 | 924 (428)
  JNJ-73763924 | 178 (73.1)

37. Secondary Outcome: Panel 2 and 3: Minimum Observed Plasma Concentration (Cmin) of JNJ-73763989 (JNJ-73763976, JNJ-73763924)
Description: Minimum observed plasma concentration (Cmin) of JNJ-73763989 (JNJ-73763976, JNJ-73763924) were reported. Non-compartmental analysis were conducted to analyze Cmin of JNJ-73763989 and its molecules
Time Frame: Week 4 (Day 29): Pre-dose and 15 minutes, 30 minutes, 1, 2, 3, 4, 6, 8, 10 and 24 hours post dose
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Panel 2 | Panel 3
Number analyzed (Participants) | 3 | 4
nanograms per milliliter (ng/mL)
  JNJ-73763976 | NA (NA) — NA indicates that mean and standard deviation were not calculable because sample concentration was below quantification limit (that is <2.1 ng/mL) | NA (NA) — NA indicates that mean and standard deviation were not calculable because sample concentration was below quantification limit (that is <2.1 ng/mL)
  JNJ-73763924 | NA (NA) — NA indicates that mean and standard deviation were not calculable because sample concentration was below quantification limit (that is <2.1 ng/mL) | NA (NA) — NA indicates that mean and standard deviation were not calculable because sample concentration was below quantification limit (that is <2.1 ng/mL)

38. Secondary Outcome: Panel 2: Time to Reach the Maximum Observed Plasma Concentration (Tmax) of JNJ-73763989 (JNJ-73763976,JNJ-73763924)
Description: Time to reach the maximum observed plasma concentration (tmax) of JNJ-73763989 (JNJ-73763976, JNJ-73763924) were reported. Non-compartmental analysis were conducted to analyze tmax of JNJ-73763989 and its molecules.
Time Frame: Week 4 (Day 29): Post dose (15 minutes, 30 minutes, 1, 2, 3, 4, 6, and 24 hours)
Population: as for outcome 35
Measure: Number; unit: hours
Arm/Group | Panel 2
Number analyzed (Participants) | 2
hours
  JNJ-73763976 - Participant 1: number analyzed (Participants) | 1
  JNJ-73763976 - Participant 1 | 6.00
  JNJ-73763976 - Participant 2: number analyzed (Participants) | 1
  JNJ-73763976 - Participant 2 | 10.00
  JNJ-73763924 - Participant 1: number analyzed (Participants) | 1
  JNJ-73763924 - Participant 1 | 6.00
  JNJ-73763924 - Participant 2: number analyzed (Participants) | 1
  JNJ-73763924 - Participant 2 | 10.00

39. Secondary Outcome: Panel 3:Time to Reach the Maximum Observed Plasma Concentration (Tmax) of JNJ-73763989 (JNJ-73763976, JNJ-73763924)
Description: as for outcome 38
Time Frame: Week 4 (Day 29): Post dose (15 minutes, 30 minutes, 1, 2, 3, 4, 6, and 24 hours)
Population: as for outcome 36
Measure: Median (Full Range); unit: hours
Arm/Group | Panel 3
Number analyzed (Participants) | 4
hours
  JNJ-73763976 | 6.00 [3.00 to 10.00]
  JNJ-73763924 | 5.04 [3.00 to 10.00]

40. Secondary Outcome: Panel 2: Area Under the Plasma Concentration-time Curve From Time Zero to 24hours (AUC0 to 24h) of JNJ-73763989 (JNJ-73763976, JNJ-73763924)
Description: Area under the plasma concentration-time curve from time zero to 24hours (AUC0 to 24h) of JNJ-73763989 (JNJ-73763976, JNJ-73763924) were reported. Non-compartmental analysis were conducted to analyze AUC0 to 24h of JNJ-73763989 and its molecules.
Time Frame: Week 4 (Day 29): Pre-dose and 15 minutes, 30 minutes, 1, 2, 3, 4, 6, 8, 10 and 24 hours post dose
Population: as for outcome 35
Measure: Number; unit: nanograms*hour per milliliters (ng*h/mL)
Arm/Group | Panel 2
Number analyzed (Participants) | 2
nanograms*hour per milliliters (ng*h/mL)
  JNJ-73763976 - Participant 1: number analyzed (Participants) | 1
  JNJ-73763976 - Participant 1 | 27744
  JNJ-73763976 - Participant 2: number analyzed (Participants) | 1
  JNJ-73763976 - Participant 2 | 13820
  JNJ-73763924 - Participant 1: number analyzed (Participants) | 1
  JNJ-73763924 - Participant 1 | 5388
  JNJ-73763924 - Participant 2: number analyzed (Participants) | 1
  JNJ-73763924 - Participant 2 | 2649

41. Secondary Outcome: Panel 3: Area Under the Plasma Concentration-time Curve From Time Zero to 24hours (AUC0 to 24h) of JNJ-73763989 (JNJ-73763976, JNJ-73763924)
Description: as for outcome 40
Time Frame: Week 4 (Day 29): Pre-dose and 15 minutes, 30 minutes, 1, 2, 3, 4, 6, 8, 10 and 24 hours post dose
Population: A pharmacokinetics (PK) analysis which included participants of Panel 3 who had consented to participate in the intensive PK subgroup. Data for this outcome measure was planned to be collected and analyzed for Panel 3 alone.
Measure: Mean (Standard Deviation); unit: nanograms*hour per milliliters (ng*h/mL)
Arm/Group | Panel 3
Number analyzed (Participants) | 4
nanograms*hour per milliliters (ng*h/mL)
  JNJ-73763976 | 13,256 (6,314)
  JNJ-73763924 | 2,394 (1,047)

ADVERSE EVENTS:
Time Frame: Open-label phase: From Day 1 (Week 1) up to Week 48; Follow-up Phase: Follow-up Week 1 up to follow-up Week 48
Description: Safety analysis set included all participants who received at least 1 dose of study intervention. Participants were analyzed according to the study intervention they actually received.
Groups:
- OL Phase: Panel 3: After PA 5, participants received either JNJ-3989 200 mg SC injection Q4W from Day 1 (Week 1) to Week 44 + JNJ-6379 250 mg QD and NA treatment (ETV 0.5 mg/TD 245 mg/TAF 25 mg) QD from Day 1 (Week 1) to Week 48, or JNJ-3989 200 mg SC injection Q4W from Day 1 (Week 1) to Week 44 + NA (ETV 0.5 mg/TD 245 mg/TAF 25 mg) QD from Day 1 (Week 1) to Week 48. After PA 5, participants discontinued JNJ-6379 and continued JNJ-3989 + NA. With separate consent, participants received optional treatment with PegIFN-alpha-2a 180 mcg SC injection QW after Week 40 liver biopsy for either 12 or 24 weeks (anytime between study Week 40 to 72) at investigator's discretion. At end of treatment Week 48, all participants entered FU phase and stopped JNJ-3989/JNJ-6379 and NA (if NA treatment completion criteria [ALT <3*ULN, HBV DNA <LLOQ; 20 IU/mL, HBeAg negative and HBsAg <10 IU/mL] was met as per Week 44 laboratory tests). If NA completion criteria were not met at Week 48, NA was continued till FU phase end (study Week 96).
- FU Phase: Panel 3: After completion of open-label study intervention phase (up to 48 weeks) all participants (HBeAg positive or negative who were either not currently treated or virologically suppressed by ETV or TD treatment) enrolled per PA 5, entered follow-up phase and stopped all study drugs (JNJ-3989 200 mg SC injection) including NA treatment [ETV 0.5 mg, TD 245 mg/TAF 25 mg], but NA treatment continued till end of follow-up (study Week 96), if NA treatment completion criteria ([ALT <3*ULN, HBV DNA <LLOQ; 20 IU/mL, HBeAg negative and HBsAg <10 IU/mL]) was not met at Week 48. Participants who were on treatment with optional PegIFN-alpha-2a 180 mcg SC injection QW after Week 40 liver biopsy but had not met NA treatment completion criteria at Week 48, were assessed at the end of treatment with PegIFN-α2a (study Week 60 or 72) and stopped NA, if the NA treatment completion criteria were met. Participants who met NA treatment completion criteria (at Week 48) were monitored Q4W in follow-up phase. If NA-retreatment criteria (HBV DNA >20,000 IU/mL, HBV DNA >2,000 IU/mL but <20,000 IU/mL & ALT >5*ULN) was met, NA retreatment was started.
Arm/Group | OL Phase: Panel 1 | OL Phase: Panel 2 | OL Phase: Panel 3 | FU Phase: Panel 1 | FU Phase: Panel 2 | FU Phase: Panel 3
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/4 | 0/10 | 0/10 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/10 | 0/4 | 0/10 | 0/10 | 0/4
Other Adverse Events (participants affected / at risk) | 9/10 | 10/10 | 3/4 | 5/10 | 6/10 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OL Phase: Panel 1 (N=10) | OL Phase: Panel 2 (N=10) | OL Phase: Panel 3 (N=4) | FU Phase: Panel 1 (N=10) | FU Phase: Panel 2 (N=10) | FU Phase: Panel 3 (N=4)
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OL Phase: Panel 1 (N=10) | OL Phase: Panel 2 (N=10) | OL Phase: Panel 3 (N=4) | FU Phase: Panel 1 (N=10) | FU Phase: Panel 2 (N=10) | FU Phase: Panel 3 (N=4)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 0 | 0
Angina Pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Eye Pruritus (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal Sounds Abnormal (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia Oral (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lip Blister (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 1 | 1 | 1 | 0 | 0 | 2
Chills (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 2 | 1 | 0 | 1 | 0
Influenza Like Illness (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Injection Site Bruising (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Injection Site Erythema (General disorders) | 1 | 1 | 0 | 0 | 0 | 0
Injection Site Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Injection Site Reaction (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 2 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Covid-19 (Infections and infestations) | 1 | 2 | 1 | 0 | 2 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0
Root Canal Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Tinea Versicolour (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0
Amylase Increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Body Temperature Increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Glomerular Filtration Rate Decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Low Density Lipoprotein Increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Weight Decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 3 | 0 | 2 | 1 | 1
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Depressed Mood (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Mood Swings (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Renal Tubular Disorder (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 2 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Rash Macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-11-25): https://cdn.clinicaltrials.gov/large-docs/89/NCT04585789/Prot_002.pdf
  • Statistical Analysis Plan (2024-02-09): https://cdn.clinicaltrials.gov/large-docs/89/NCT04585789/SAP_003.pdf